CLINICAL TRIAL: NCT00936663
Title: A Randomized, Placebo-Controlled Double-Blind Trial Using Sitagliptin as a Treatment to Prevent New Onset Diabetes After Kidney Transplantation: A Pilot Study
Brief Title: Using Sitagliptin as a Treatment to Prevent New Onset Diabetes After Kidney Transplantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0254-09-FB
Record Dates: First submitted 2009-06-25; First posted 2009-07-10 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: Type 2 Diabetes; End Stage Renal Disease
Keywords: Diabetes; Kidney Transplant; Sitagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Kidney Failure, Chronic; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin 100 mg daily (Experimental): sitagliptin 100 mg daily
  Interventions: Drug: Sitagliptin
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Active drug dose will be 100 mg per day for estimated GFR above 50 ml/min. The dose will be decreased to 50 mg per day for estimated GFR 30-50 ml/min. The dose will be decreased further to 25 mg for those with estimated GFR below 30 ml/min or on dialysis.
  Arms: placebo
Drug: Sitagliptin — Active drug dose will be 100 mg per day for estimated GFR above 50 ml/min. The dose will be decreased to 50 mg per day for estimated GFR 30-50 ml/min. The dose will be decreased further to 25 mg for those with estimated GFR below 30 ml/min or on dialysis.
  Arms: Sitagliptin 100 mg daily

SUMMARY:
This study is designed to see if the use of the drug Sitagliptin (used to reduce insulin resistance) will delay or prevent kidney transplant patients from getting diabetes.

DETAILED DESCRIPTION:
New-onset diabetes after transplantation (NODAT) is a complication of solid organ transplantation. In the University of Nebraska Medical Center (UNMC) Kidney-Pancreas Transplant Clinic, the frequency of this complication exceeds 50% of kidney transplant recipients without diabetes prior to transplantation. NODAT is associated with increased morbidity and mortality. As this complication appears to occur rather soon after transplantation, potential preventative strategies need to be instituted soon after transplantation. Although traditional risk factors, such as family history, obesity, and minority status, explain some of the additional risk, it is thought that the immunosuppressive agents themselves are responsible for the increased risk of NODAT. The immunosuppressive agents are needed to prevent rejection, and we are left to consider additional strategies to prevent the onset of NODAT. This is a pilot study utilizing the dipeptidyl peptidase-4 inhibitor, sitagliptin, in a randomized, double-blinded, placebo-controlled study in consecutive kidney transplant recipients at the University of Nebraska Medical Center. Sitagliptin has been tested in patients with type 2 diabetes who have received a kidney transplant and have shown no major side effects or alterations in immunosuppressive drug levels. This agent is FDA-approved for the treatment of type 2 diabetes, but it has a low rate of hypoglycemia. It is thought to work by inhibiting the enzyme that naturally breaks down glucagons-like peptide-1 (GLP-1), thus increasing endogenous levels of GLP-1. GLP-1 inhibits glucagons and has stimulatory effects on beta cell function. Although the current study will treat all non-diabetic patients in the hope that NODAT is delayed or prevented, this incretin-based therapy is thought to have a low risk for hypoglycemia and other side effects. In addition, it can be safely used during low-GFR conditions. The study will attempt to recruit 40 subjects (20 sitagliptin and 20 control subjects). Patients will initiate placebo or control at 2 weeks after transplantation. Subjects will be followed in the UNMC Transplant Clinic. Initially, patients will be seen weekly and later will be followed every three months for up to 1 year. The primary outcome is the development of NODAT based on the 2003 Consensus International Guidelines. Fasting glucose levels will be followed according to usual post-transplant monitoring with testing as frequently as weekly during the recent post-transplant period and eventually going to at least monthly. Secondary outcomes include HbA1c values and glucose, insulin, C-peptide, and proinsulin levels after a 75 oral glucose load that will be obtained at baseline and then every three months. In addition, side effects, including hypoglycemia, will be followed. The study will have a local Data Safety Monitoring Board (DSMB). Consent will be obtained prior to transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Recipient of a kidney transplant at UNMC, including cadaveric or living donor transplant.

Exclusion Criteria:

* A previous diagnosis of diabetes or previous criteria for diabetes, according to the American Diabetes Association, not previously recognized as diabetes.
* Simultaneous transplant of another solid organ, such liver or heart.
* Patient unable to take oral medication.
* Patient unable to give informed consent.
* Hypersensitivity to sitagliptin.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-07-06 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2010-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Shivaswamy, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Background] Lane JT, Odegaard DE, Haire CE, Collier DS, Wrenshall LE, Stevens RB. Sitagliptin therapy in kidney transplant recipients with new-onset diabetes after transplantation. Transplantation. 2011 Nov 27;92(10):e56-7. doi: 10.1097/TP.0b013e3182347ea4. No abstract available. PMID 22067216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: 10/2009 to 8/2012 Recruitment location: Transplant Clinic and Nebraska Medicine Hospital
Pre-assignment Details: 1 subject consented, but dropped out as she was too busy to participate in the study
Period: Overall Study
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg Daily | Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (0) | 34 (9.9) | 41 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3
HbA1c [Mean (Standard Deviation); unit: percentage of glycated haemoglobin] | 5.6 (0) | 5.8 (1.5) | 5.7 (1.0)
Fasting Blood Glucose [Mean (Standard Deviation); unit: mg/dl] | 105 (0) | 125 (25.5) | 118.3 (21.3)
estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m²] | 48 (0) | 32 (9.9) | 37.3 (11.6)
Area Under the Curve (AUC) for glucose [Mean (Standard Deviation); unit: mg*hr/dl] — Population: Baseline OGTT was not performed in one patient in Sitagliptin group and one patient in placebo group
  Reason was not documented
  mg*hr/dl
    number analyzed (Participants) | 0 | 1 | 1
    (all) |  | 408 (0) | 408 (0)
AUC for Insulin [Mean (Standard Deviation); unit: mciu*hr/ml] — Population: Baseline OGTT was not performed in one patient in Sitagliptin group and one patient in placebo group Reason was not documented
  mciu*hr/ml
    number analyzed (Participants) | 0 | 1 | 1
    (all) |  | 101.5 (0) | 101.5 (0)
AUC Proinsulin [Mean (Standard Deviation); unit: pmol*hr/L] — Population: Baseline OGTT was not performed in one patient in Sitagliptin group and one patient in placebo group Reason was not documented
  pmol*hr/L
    number analyzed (Participants) | 0 | 1 | 1
    (all) |  | 52.5 (0) | 52.5 (0)
AUC C peptide [Mean (Standard Deviation); unit: ng*hr/ml] — Population: Baseline OGTT was not performed in one patient in Sitagliptin group and one patient in placebo group Reason was not documented
  ng*hr/ml
    number analyzed (Participants) | 0 | 1 | 1
    (all) |  | 26.8 (0) | 26.8 (0)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Blood Glucose
Description: Fasting blood glucose levels at 1 year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Number analyzed (Participants) | 1 | 2
mg/dl | 107 (0) | 102.5 (7.8)

2. Secondary Outcome: HbA1c
Description: HbA1c at 1 year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: percentage of glycated haemoglobin
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Number analyzed (Participants) | 1 | 2
percentage of glycated haemoglobin | 6.1 (0) | 5.8 (0.9)

3. Secondary Outcome: eGFR
Description: estimated glomerular filtration rate (eGFR) at 1 year
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m²
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Number analyzed (Participants) | 1 | 2
mL/min/1.73 m² | 52 (0) | 41.5 (16.3)

4. Secondary Outcome: Hypoglycemia
Description: Number of episodes of hypoglycemia (blood glucose less than 70 mg/dl)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Number analyzed (Participants) | 1 | 2
episodes | 0 (0) | 0 (0)

5. Other Pre Specified Outcome: AUC for Glucose
Description: Area Under the Curve for glucose after OGTT
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mg*hr/dl
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Number analyzed (Participants) | 1 | 2
mg*hr/dl | 277.5 (0) | 336.5 (101.1)

6. Other Pre Specified Outcome: AUC for Insulin
Description: Area Under the Curve for insulin after OGTT
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mciu*hr/ml
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Number analyzed (Participants) | 1 | 2
mciu*hr/ml | 72.5 (0) | 85.75 (5.3)

7. Other Pre Specified Outcome: AUC for Proinsulin
Description: Area Under the Curve for Proinsulin after OGTT
Time Frame: 1 year
Measure: Mean (Standard Error); unit: pmol*hr/L
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Number analyzed (Participants) | 1 | 2
pmol*hr/L | 62.6 (0) | 44.83 (39.14)

8. Other Pre Specified Outcome: AUC for C Peptide
Description: Area Under the Curve for C peptide after OGTT
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | Sitagliptin 100 mg Daily | Placebo
Number analyzed (Participants) | 1 | 2
ng*hr/ml | 19.5 (0) | 23.28 (16.65)

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Sitagliptin 100 mg Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 100 mg Daily (N=1) | Placebo (N=2)
Non-Fatal Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Acute anterior wall myocardial infarction on January 29, 2012. Patient has chronic kidney disease, long standing hypertension and anemia which are known risk factors for cardiovascular disease.

LIMITATIONS AND CAVEATS:
We did not reach the target number of participants needed to achieve target power and statistically reliable results as the funding was not renewed by the sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No